CLINICAL TRIAL: NCT07228585
Title: Comparison of the Effects of Kinesio Taping and Interval Exercise in Patients Diagnosed With Venous Insufficiency: A Randomised Controlled Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Enise Neval Arslan, Physiotherapist (MSc student in Physiotherapy and Rehabilitation), Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 25936
Record Dates: First submitted 2025-11-13; First posted 2025-11-14 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Chronic Venous Insufficiency C2 and Below
Keywords: venous insufficiency; kinesiology tape; interval training; lifestyle recommendations; physiotherapy and rehabilitation; physiotherapy
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Intervention Model Description: The interventional study model evaluates the effects of specific treatments on defined groups. It actively applies an intervention and measures outcomes such as symptoms, function, or quality of life. Randomization assigns participants to experimental or control groups to reduce bias, ensuring observed effects are due to the intervention. In physiotherapy, interventions may include exercise, taping, or manual therapy, with outcomes assessed before and after treatment. Ethical approval, informed consent, and standardized procedures are essential. Despite resource demands, this model provides reliable evidence, guiding clinical decisions and improving patient outcomes.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Active Comparator: KT + Advice (Active Comparator): Participants receive lifestyle modification advice for venous insufficiency, including reducing prolonged standing, interrupting sitting with leg movements, and elevating legs above heart level. All participants are advised on daily physical activity (at least 30 minutes of brisk walking), leg elevation (2-3 times for 15-20 minutes), low-salt and high-fiber diet, hydration, smoking cessation, and skin care. Kinesio taping is applied using lymphatic correction techniques from the popliteal area to the lower leg (15-20% tension), changed twice weekly for eight weeks.
  Interventions: Behavioral: Kinesio Taping and Lifestyle Advice
- Experimental: KT + Exercise + Advice (Experimental): Participants receive standard lifestyle advice as described for venous insufficiency and Kinesio taping using lymphatic correction techniques (popliteal to lower leg, covering gastrocnemius, soleus, and tibialis posterior, 15-20% tension). Tape is replaced twice weekly for eight weeks. Interval exercise is performed three times weekly for 30-40 minutes, consisting of warm-up, alternating low- and moderate-intensity phases, and cool-down with stretching and diaphragmatic breathing. Weekly monitoring ensures safety and adherence.
  Interventions: Behavioral: Kinesio Taping and Interval Exercise with Lifestyle Advice
- Active Comparator: Advice Only (Active Comparator): Participants receive comprehensive lifestyle modification advice for venous insufficiency, including reduction of prolonged standing, frequent leg movements, leg elevation above heart level, regular physical activity, low-salt and high-fiber diet, hydration, smoking cessation, suitable clothing, and skin moisturizing. All guidance is delivered by physiotherapists, considering individual medical history and contraindications
  Interventions: Behavioral: Lifestyle Advice for Venous Insufficiency

INTERVENTIONS:
Behavioral: Kinesio Taping and Lifestyle Advice — Participants receive lifestyle modification advice for venous insufficiency, including reducing prolonged standing, interrupting sitting with leg movements, and elevating legs above heart level. All participants are advised on daily physical activity (at least 30 minutes of brisk walking), leg elevation (2-3 times for 15-20 minutes), low-salt and high-fiber diet, hydration, smoking cessation, and skin care. Kinesio taping is applied using lymphatic correction techniques from the popliteal area to the lower leg (15-20% tension), changed twice weekly for eight weeks.
  Arms: Active Comparator: KT + Advice
Behavioral: Kinesio Taping and Interval Exercise with Lifestyle Advice — Participants receive standard lifestyle advice as described for venous insufficiency and Kinesio taping using lymphatic correction techniques (popliteal to lower leg, covering gastrocnemius, soleus, and tibialis posterior, 15-20% tension). Tape is replaced twice weekly for eight weeks. Interval exercise is performed three times weekly for 30-40 minutes, consisting of warm-up, alternating low- and moderate-intensity phases, and cool-down with stretching and diaphragmatic breathing. Weekly monitoring ensures safety and adherence.
  Arms: Experimental: KT + Exercise + Advice
Behavioral: Lifestyle Advice for Venous Insufficiency — Participants receive comprehensive lifestyle modification advice for venous insufficiency, including reduction of prolonged standing, frequent leg movements, leg elevation above heart level, regular physical activity, low-salt and high-fiber diet, hydration, smoking cessation, suitable clothing, and skin moisturizing. All guidance is delivered by physiotherapists, considering individual medical history and contraindications.
  Arms: Active Comparator: Advice Only

SUMMARY:
This study aims to compare the effects of kinesiology taping and interval exercise on reducing symptoms, improving quality of life, and vital parameters in individuals with venous insufficiency. The study will be conducted at the Department of Cardiovascular Surgery, Faculty of Medicine, Necmettin Erbakan University, Konya, and will involve individuals aged 18 to 65 who have been diagnosed with venous insufficiency. Participants will be selected according to inclusion criteria and randomised into three groups. These groups will consist of a group receiving kinesiology taping and lifestyle recommendations, a group receiving kinesiology taping combined with interval exercise and lifestyle recommendations, and a control group receiving only lifestyle recommendations. Participants will be followed up for eight weeks, with assessments conducted twice: before and after treatment.

In kinesiology taping groups, taping will be applied twice a week for eight weeks, with a total of sixteen sessions. During application, the lymphatic correction technique will be used to increase venous circulation. Taping will begin over the popliteal vein and be applied along the gastrocnemius, soleus, and tibialis posterior muscles with a tension of fifteen to twenty per cent. Participants will inform the physiotherapist if they experience any discomfort or skin sensitivity related to the bandaging, and skin reactions and tolerance levels will be monitored during weekly check-ups. In the group undergoing interval exercise, participants will participate in a mild to moderate exercise programme for thirty to forty minutes, three days a week for eight weeks. The exercises will be performed under the supervision of a physiotherapist and will be of an intensity equivalent to levels three to five on the Borg scale. The programme will include a five-minute warm-up phase, a twenty-minute main exercise section, and a five-minute cool-down period. The main section will consist of three phases, with low-intensity, moderate-intensity, and recovery exercises applied alternately. In the low-intensity section, light-paced walking and step movements will be performed; in the moderate-intensity section, fast-paced walking, ankle pumping movements, squats or calf raises will be performed; in the recovery section, light walking or wrist movements will be preferred. The main exercise will be completed after the cycle is repeated four times, followed by light stretching movements and diaphragmatic breathing exercises during the cool-down phase. Exercise compliance will be monitored on a weekly basis.

Standard lifestyle recommendations will be provided to all groups participating in the study. As lifestyle changes in venous insufficiency have both therapeutic and symptom-reducing effects, participants will be given detailed information on this subject. Lifestyle recommendations include increasing physical activity habits such as walking briskly for at least thirty minutes daily and using stairs. As part of leg elevation recommendations, it will be advised to keep the legs above heart level for fifteen to twenty minutes, two or three times a day. Individuals whose jobs require them to stand still for long periods will be advised to take a short walk every thirty minutes. Nutritional recommendations will emphasise reducing salt intake, drinking at least two litres of water daily, and eating fibre-rich foods. Smoking participants will be counselled to quit and asked to avoid wearing tight trousers and high-heeled shoes. As part of skin care, participants will be instructed to use moisturiser once a day to prevent dryness and cracking in the lower extremities. Lifestyle recommendations will be presented to participants via a brochure, and participants in the control group will also follow the same recommendations.

The conditions of the study and safety measures have been determined with great care. All procedures will be performed by experienced physiotherapists, taking into account the participants' medical history and contraindications. Assessments will be conducted twice: at the beginning and at the end of the eight-week period. Measurements will include ankle circumference, pain intensity at rest, during sleep and during exercise, blood pressure, heart rate, respiratory rate, body temperature, oxygen saturation, Borg scale assessment, physical activity level measurement, functional capacity assessment, central sensitisation level and quality of life in venous insufficiency. The six-minute walk test will be used to assess functional capacity, the visual analogue scale will be applied for pain, this parameter will be examined using the central sensitisation inventory, and quality of life will be assessed using scales specific to venous insufficiency. The International Physical Activity Questionnaire will be used for physical activity level.

DETAILED DESCRIPTION:
Inclusion criteria for the study include being aged between 18 and 65, having a diagnosis of chronic venous insufficiency, being in stages 0 to 2 of the CEAP classification, having no health problems that would prevent participation in physical activity, being able to read and understand Turkish, and having no allergy to kinesiology taping. Exclusion criteria from the study were defined as having a diagnosis of acute venous thrombosis, a history of serious cardiovascular disease, pregnancy or breastfeeding, the presence of an active infection, and unwillingness to continue participating in the study.

The data collection process will be conducted through face-to-face interviews and observation methods. Participants' demographic and clinical information will be obtained from patient files, and measurements will be taken using specified scales and tests. All data will be recorded by researchers and protected in accordance with confidentiality principles. Participants' identity information will not be included in the records; each participant will be assigned a unique code number. Data will be stored in an encrypted digital environment accessible only to the researcher and will not be shared with third parties. Identity information will be completely anonymised in the study reports. Written informed consent will be obtained from all participants before the study begins. The study will be conducted in accordance with the Declaration of Helsinki.

The three distinct groups established within this research will enable the assessment of both treatment efficacy and its impact on quality of life. Kinesiology taping aims to reduce oedema and symptoms by enhancing lymphatic flow and venous return. Interval exercises are employed to strengthen circulation, activate the muscle pump, and increase functional capacity. Lifestyle recommendations will support symptom relief through small changes in individuals' daily lives, while forming a standard basis across all groups. The data obtained from the study will enable a scientific comparison of the effectiveness of different approaches in the treatment of venous insufficiency, with a particular focus on evaluating the contribution of combined exercise and taping applications.

Ultimately, this research aims to provide important findings that will guide clinical practice by enabling the comparison of different treatment approaches in individuals with venous insufficiency. Examining the effects of kinesiology taping and interval exercise on quality of life, functional capacity, symptom severity, and vital parameters will both increase patient compliance with treatment and provide physiotherapists with a scientific basis for their practice.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 18-65
* Individuals diagnosed with chronic venous insufficiency (those in stages 0-2 of the CEAP classification)
* Individuals with no barriers to participating in physical activity
* Individuals who can read and understand Turkish and have no communication difficulties
* Individuals with no allergy to kinesiology taping in the kinesiology taping group

Exclusion Criteria:

* Diagnosis of acute venous thrombosis
* History of serious cardiovascular disease
* Pregnancy or breastfeeding
* Presence of active infection
* Those who do not wish to continue participating in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-02-08 (Actual); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in Central Sensitization Inventory (CSI Part A Score) | At baseline (before intervention) and after 8 weeks of intervention.
  Central sensitization symptoms will be assessed using the Central Sensitization Inventory (CSI) Part A. Total score ranges from 0 to 100, with higher scores indicating greater central sensitization.
  Time Frame: At baseline (before intervention) and after 8 weeks of intervention.

SECONDARY OUTCOMES:
Change in Central Sensitization Inventory (CSI Part B) | At baseline (before intervention) and after 8 weeks of intervention.
  The number of clinician-diagnosed central sensitivity syndromes will be documented using the Central Sensitization Inventory (CSI) Part B.
  Time Frame: At baseline (before intervention) and after 8 weeks of intervention.
Change in Venous Insufficiency-Specific Quality of Life (VEINES-QOL/Sym) | At baseline (before intervention) and after 8 weeks of intervention.
  Quality of life and symptom severity will be evaluated using the VEINES-QOL/Sym questionnaire. Higher scores indicate better quality of life and fewer venous symptoms.
  Time Frame: At baseline (before intervention) and after 8 weeks of intervention.
Change in Pain Intensity (Visual Analog Scale, VAS) | At baseline (before intervention) and after 8 weeks of intervention.
  Pain intensity at rest and during activity will be measured using the Visual Analog Scale (VAS), ranging from 0 (no pain) to 10 (worst imaginable pain).
  Time Frame: At baseline (before intervention) and after 8 weeks of intervention.
Change in Functional Capacity (6-Minute Walk Test) | At baseline (before intervention) and after 8 weeks of intervention.
  Functional capacity will be assessed using the 6-Minute Walk Test. The total distance (in meters) covered during 6 minutes will be recorded.
Change in Perceived Exertion (Modified Borg Scale) | At baseline (before intervention) and after 8 weeks of intervention.
  Perceived exertion during exercise will be evaluated using the Modified Borg Scale (0-10). Higher scores indicate greater exertion.
Change in Physical Activity Level (International Physical Activity Questionnaire, IPAQ) | At baseline (before intervention) and after 8 weeks of intervention.
  Physical activity level will be assessed using the short form of the International Physical Activity Questionnaire (IPAQ). Results will be expressed in MET-minutes per week.

CONTACTS AND LOCATIONS:
Locations (1):
- Necmettin Erbakan University, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The Individual Participant Data (IPD) Sharing Plan is confirmed as "Yes." All de-identified participant-level data collected during the study-including clinical measurements, assessments, and outcome data forming the basis of the study's publications-will be shared. Data will be made available upon reasonable request for secondary analyses, replication studies, or meta-analyses. All data sharing will adhere to strict confidentiality protocols to protect participant privacy, ensuring that no identifiable information is disclosed. Access procedures, including necessary approvals and data use agreements, will be established to facilitate secure and responsible data dissemination.
Supporting Information: Study Protocol, SAP, ICF, CSR